CLINICAL TRIAL: NCT01784120
Title: A Phase II Trial of Doxorubicin and Genexol-PM in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyung Cho, Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-GIRBA-2566
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; doxorubicin; genexol-PM; paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; genexol-PM

ARMS (1):
- doxotubicin/Genexol-PM (Experimental)
  Interventions: Drug: Doxorubicin/Genexol-PM

INTERVENTIONS:
Drug: Doxorubicin/Genexol-PM

SUMMARY:
To evaluate efficacy and toxicity of doxorubicin/Genexol-PM in metastatic breast cancer

1. Primary Purpose: response rate
2. Secondary purpose: toxicity, progression-free survival, overall survival

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older adult women
* Instrumentation measurable lesions with histologically confirmed advanced (recurrent or metastatic) breast cancer
* ECOG 0-2
* Advanced breast cancer in the past, patients who did not receive chemotherapy
* Recurrence if adjuvant chemotherapy and adjuvant chemotherapy in the past for more than 6 months until the patient
* life expectancy more than 3 months
* Agree in writing before the party to participate in a clinical trial to patients

Exclusion Criteria:

* immunohistochemical staining 3 + or FISH positive anti-HER 2 therapy patients
* Severe infections requiring antibiotic therapy
* Clinically significant heart disease
* Pregnant or lactating woman
* Uncontrolled symptoms in the central nervous system (CNS) metastases
* Patients diagnosed with malignant tumors of other organs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
response rate | one year

SECONDARY OUTCOMES:
number of participants with adverse events | one year

OTHER OUTCOMES:
overall survival | one year
progression-free-survival | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea